CLINICAL TRIAL: NCT03850535
Title: A Phase Ib/II Study Evaluating the Safety and Efficacy of Idasanutlin in Combination With Cytarabine and Daunorubicin in Patients Newly Diagnosed With Acute Myeloid Leukemia (AML) and the Safety and Efficacy of Idasanutlin in the Maintenance of First AML Complete Remission
Brief Title: A Study Evaluating the Safety and Efficacy of Idasanutlin in Combination With Cytarabine and Daunorubicin in Patients Newly Diagnosed With Acute Myeloid Leukemia (AML) and the Safety and Efficacy of Idasanutlin in the Maintenance of First AML Complete Remission
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision to terminate the study after Phase 1; will not proceed with Phase 2.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO40800; 2018-002964-25 (EudraCT Number)
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Results first posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — RG7388; Cytarabine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose-Escalation Phase (Experimental): Participants with newly diagnosed, previously untreated, favorable or intermediate risk AML (according to European LeukemiaNet [ELN] 2017 criteria) will undergo the treatment sequence of induction, consolidation, and maintenance. For induction, participants will be treated with idasanutlin plus cytarabine and daunorubicin. At the investigator's discretion for consolidation, either participants will be treated with idasanutlin and cytarabine or they will undergo Allo-HSCT. For maintenance, participants will be treated with single-agent idasanutlin.
  Interventions: Drug: Idasanutlin; Drug: Cytarabine; Drug: Daunorubicin; Procedure: Allogeneic Hematopoietic Stem Cell Transplant (Allo-HSCT)
- Post-Consolidation Phase (Experimental): Participants who are idasanutlin treatment-naive, had received induction and chemotherapy consolidation for AML outside of the study, and were in minimal residual disease (MRD)-positive remission after induction will be enrolled in this cohort to receive maintenance treatment with single-agent idasanutlin.
  Interventions: Drug: Idasanutlin
- Expansion Phase: Favorable/Intermediate-Risk AML (Experimental): Participants with newly diagnosed, previously untreated, favorable or intermediate risk AML (according to ELN 2017 criteria) will undergo the treatment sequence of induction, consolidation, and maintenance. For induction, participants will be treated with idasanutlin (at the recommended Phase 2 dose) plus cytarabine and daunorubicin. At the investigator's discretion for consolidation, either participants will be treated with idasanutlin and cytarabine or they will undergo Allo-HSCT. For maintenance, participants will be treated with single-agent idasanutlin.
  Interventions: Drug: Idasanutlin; Drug: Cytarabine; Drug: Daunorubicin; Procedure: Allogeneic Hematopoietic Stem Cell Transplant (Allo-HSCT)
- Expansion Phase: High-Risk AML (Experimental): Participants with newly diagnosed, previously untreated, high-risk AML (defined as adverse risk according to ELN 2017 criteria, and secondary AML) will undergo the treatment sequence of induction, consolidation, and maintenance. For induction, participants will be treated with idasanutlin (at the recommended Phase 2 dose) plus cytarabine and daunorubicin. At the investigator's discretion for consolidation, either participants will be treated with idasanutlin and cytarabine or they will undergo Allo-HSCT. For maintenance, participants will be treated with single-agent idasanutlin.
  Interventions: Drug: Idasanutlin; Drug: Cytarabine; Drug: Daunorubicin; Procedure: Allogeneic Hematopoietic Stem Cell Transplant (Allo-HSCT)

INTERVENTIONS:
Drug: Idasanutlin — Participants will self-administer idasanutlin tablets by mouth (PO) once daily (QD) for 5 days of each 28-day treatment cycle for up to 2 cycles of induction, up to 4 cycles of consolidation, and 12 cycles of maintenance, according to the study's protocol.
  Other Names: RO5503781; RG7388
Drug: Cytarabine — Cytarabine will be administered for 7 days of each 28-day cycle for up to 2 cycles of induction treatment at a dose of 200 milligrams per meter squared (mg/m^2) of body surface area, once daily (QD) by intravenous (IV) infusion. At the investigator's discretion, cytarabine will also be administered as part of chemotherapy consolidation at a dose of 1.5 g/m^2 QD as IV infusion for 5 days of each 28-day cycle and for up to 4 cycles of treatment.
  Arms: Dose-Escalation Phase; Expansion Phase: Favorable/Intermediate-Risk AML; Expansion Phase: High-Risk AML
Drug: Daunorubicin — Daunorubicin will be administered for 3 days of each 28-day cycle for up to 2 cycles of induction treatment at a dose of 60 mg/m^2 QD as IV infusion.
  Arms: Dose-Escalation Phase; Expansion Phase: Favorable/Intermediate-Risk AML; Expansion Phase: High-Risk AML
Procedure: Allogeneic Hematopoietic Stem Cell Transplant (Allo-HSCT) — After induction treatment, participants who achieve remission will either receive chemotherapy consolidation treatment or undergo Allo-HSCT (as per local guidelines) at the investigator's discretion.
  Arms: Dose-Escalation Phase; Expansion Phase: Favorable/Intermediate-Risk AML; Expansion Phase: High-Risk AML

SUMMARY:
This Phase Ib/II, open-label, multicenter, non-randomized study will evaluate the safety, efficacy, and pharmacokinetics of idasanutlin when it is given in combination with cytarabine and daunorubicin in induction, in combination with cytarabine in consolidation, and as a single agent in maintenance for treating participants with acute myeloid leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for All Study Phases:

* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Adequate hepatic and renal function
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating eggs with a failure rate of <1% per year during the treatment period and for at least 6 months after the final dose of idasanutlin, cytarabine, or daunorubicin. Women must refrain from donating eggs during this same period.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive, measures, and agreement to refrain from donating sperm that together result in a failure rate of <1% per year during the treatment period and for 6 months after the final dose of idasanutlin, cytarabine, or daunorubicin. Men must refrain from donating sperm during this same period.

Inclusion Criteria for Patients in the Dose-Escalation and Expansion Phases:

- Documented/confirmed newly diagnosed acute myeloid leukemia (AML) not previously treated according to World Health Organization (WHO)

Inclusion Criteria for Patients in the Post-Consolidation Phase:

- Documented/confirmed AML according to WHO in remission after induction, within 21 days of end of last chemotherapy consolidation cycle, and were minimum residual disease (MRD) positive at the end of induction as per local laboratory assessment

Exclusion Criteria:

Exclusion Criteria for All Study Phases:

* Clinical evidence of central nervous system (CNS) leukemia
* Any Grade ≥2 non-hematologic toxicities prior to starting therapy
* Current treatment with any other investigational or commercial agents or therapies administered with the intention to treat their malignancy with the exception of hydroxyurea (HU) or 6-mercaptopurine (6-MP)
* Treatment-related AML
* Acute promyelocytic leukemia
* History of other malignancy that could affect compliance with the protocol or interpretation of results
* Any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study, impair the ability of the investigator to evaluate the patient, or impair the patient's ability to complete the study
* Echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan showing ejection fraction ≤40%
* Non-malignant medical illnesses that are uncontrolled or whose control may be jeopardized by this study treatment, such as hereditary coagulation disorders, insulin-dependent diabetes mellitus not optimally controlled with medical management (e.g., presence of ketoacidosis), or active GI conditions affecting absorption
* Infection considered by the investigator to be clinically uncontrolled or of unacceptable risk to the patient upon the induction of neutropenia, that is, patients who are or should be on antimicrobial agents for the treatment of active infection
* Febrile patients within 72 hours of study treatment initiation
* Patients with a history of active or chronic infectious hepatitis unless serology demonstrates clearance of infection
* Patients who are unable to interrupt treatment with moderate to strong CYP2C8 inducers and inhibitors
* Patients who are unable to temporarily interrupt treatment with oral or parenteral anticoagulants/anti-platelet agents during treatment phase
* Patients who have a history of clinically significant liver cirrhosis
* Patients with extramedullary AML with no evidence of systemic involvement
* Pregnant or breastfeeding patients
* Known history of HIV-positive status
* Patients who might refuse to receive blood products and/or have a hypersensitivity to blood products
* Prior treatment with an MDM2 antagonist
* Patients with clinically relevant QTc prolongation, a family history of long QT syndrome

Exclusion Criteria for Patients in the Phase Ib Dose-Escalation Phase:

- Adverse risk patients as per European LeukemiaNet (ELN) 2017 criteria

Exclusion Criteria for Patients in Phase Ib Post-Consolidation Phase:

* Any ongoing Grade ≥2 hematologic adverse events prior to starting therapy
* Previous hematopoietic stem cell transplant (HSCT)

Exclusion Criteria for Patients in the Dose-Escalation Phase and Patients in the Favorable/Intermediate-Risk Cohort of the Expansion Phase:

- Secondary AML, defined as AML evolving from antecedent hematologic disorder (AHD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- United States (12):
  - UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - University of Iowa Hospitals and Clinics; Investigational Drug Services, Iowa City, Iowa
  - University of Kansas Clinical Research Center; Clinical Trials Office, Fairway, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - State University of NY, Brooklyn, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - The Alfred Hospital, Prahan, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- France (5):
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHU de Nantes - Hotel Dieu, Nantes
  - Hôpital Saint-Louis, Paris
  - Institut Universitaire du Cancer de Toulouse-Oncopole, Toulouse
- Italy (2):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST); Onco-Ematologia, Meldola, Emilia-Romagna
  - ASST Papa Giovanni XXIII; Dipartimento Interaziendale di Farmacia Clinica, Bergamo, Lombardy
- Spain (5):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz., Madrid
  - Hospital Universitario Virgen del Rocío; Servicio de Neuropediatra, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose-Escalation Cohort 1: 200 mg idasanutlin day 1 to day 5 in combination with cytarabine 200mg day 1 to day 7 and daunorubicin 60mg day 1 to day 3 in induction
- Dose Escalation Cohort 2: 350 mg idasanutlin day 1 to day 5 in combination with cytarabine 200mg day 1 to day 7 and daunorubicin 60mg day 1 to day 3 in induction
- Dose Escalation Cohort 3: 250 mg idasanutlin day 1 to day 5 in combination with cytarabine 200mg day 1 to day 7 and daunorubicin 60mg day 1 to day 3 in induction
- Post Consolidation Cohort: 150 mg idasanultin day 1 to 5 in maintenance of first remission
Period: Overall Study
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Started | 4 | 9 | 6 | 4
Completed | 0 | 0 | 0 | 0
Not Completed | 4 | 9 | 6 | 4

BASELINE CHARACTERISTICS:
Population: There was no expansion phase taken place.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort | Total
Number analyzed (Participants) | 4 | 9 | 6 | 4 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.5 (17.1) | 45.2 (16.9) | 49.8 (14.0) | 64.8 (7.2) | 50.6 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 3 | 11
  Male | 2 | 6 | 3 | 1 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 5 | 0 | 6
  Not Hispanic or Latino | 2 | 9 | 0 | 3 | 14
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 3 | 7 | 4 | 3 | 17
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation Phase: Number of Participants With Dose-Limiting Toxicities (DLTs) During the First Cycle of Induction Treatment
Description: Sponsor's decision to prematurely terminate the study was made at the end of the Phase 1. The planned Phase 2 was not initiated. This decision was not based on safety concerns, but rather due to the overall company strategy about the adult AML
Time Frame: Cycle 1 of induction treatment (1 cycle is 28 days)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 4 | 9 | 6 | 4
Participants | 2 | 4 | 0 | 0

2. Primary Outcome: Number of Participants With at Least One Adverse Event
Description: as for outcome 1
Time Frame: From Baseline until 28 days after the final dose of study drug (up to 2 years)
Population: Safety Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 4 | 9 | 6 | 4
Percentage of Participants | 4 | 9 | 6 | 4

3. Primary Outcome: Number of Participants With Grade ≥3 Adverse Events, Severity Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)
Description: as for outcome 1
Time Frame: From Baseline until 28 days after the final dose of study drug (up to 2 years)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 4 | 9 | 6 | 4
Participants | 4 | 9 | 5 | 4

4. Primary Outcome: Number of Participants Reporting Presence or Absence of Nausea Over Time, as Assessed Through Use of the National Cancer Institute (NCI) Patient-Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Description: The sponsor decided not to continue the study based on the overall Company strategy in AML. Although data were collected, the small sample size and insufficient follow up rendered any analysis scientifically meaningless. As a consequence, no data were analyzed and this outcome measure was not conducted
Time Frame: Day 1 of each treatment cycle (1 cycle is 28 days) and at study drug discontinuation (up to 2 years)
Population: Due to the insufficient enrollment of the planned Analysis Population, the planned outcome measurements were not conducted and result data were not collected.
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Primary Outcome: Change From Baseline Over Time in Reported Frequency of Nausea, as Assessed Through Use of the NCI PRO-CTCAE
Description: as for outcome 4
Time Frame: Baseline, Day 1 of each treatment cycle (1 cycle is 28 days), and at study drug discontinuation (up to 2 years)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Primary Outcome: Change From Baseline Over Time in Reported Severity of Nausea, as Assessed Through Use of the NCI PRO-CTCAE
Description: as for outcome 4
Time Frame: Baseline, Day 1 of each treatment cycle (1 cycle is 28 days), and at study drug discontinuation (up to 2 years)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Primary Outcome: Change From Baseline Over Time in Reported Degree of Interference With Daily Function Caused by Nausea, as Assessed Through Use of the NCI PRO-CTCAE
Description: as for outcome 4
Time Frame: Baseline, Day 1 of each treatment cycle (1 cycle is 28 days), and at study drug discontinuation (up to 2 years)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Primary Outcome: Change From Baseline Over Time in Overall Score for Nausea, as Assessed Through Use of the NCI PRO-CTCAE
Description: as for outcome 4
Time Frame: Baseline, Day 1 of each treatment cycle (1 cycle is 28 days), and at study drug discontinuation (up to 2 years)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants Reporting Presence or Absence of Vomiting Over Time, as Assessed Through Use of the NCI PRO-CTCAE
Description: as for outcome 4
Time Frame: Day 1 of each treatment cycle (1 cycle is 28 days) and at study drug discontinuation (up to 2 years)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Primary Outcome: Change From Baseline Over Time in Reported Frequency of Vomiting, as Assessed Through Use of the NCI PRO-CTCAE
Description: as for outcome 4
Time Frame: Baseline, Day 1 of each treatment cycle (1 cycle is 28 days), and at study drug discontinuation (up to 2 years)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Primary Outcome: Change From Baseline Over Time in Reported Severity of Vomiting, as Assessed Through Use of the NCI PRO-CTCAE
Description: as for outcome 4
Time Frame: Baseline, Day 1 of each treatment cycle (1 cycle is 28 days), and at study drug discontinuation (up to 2 years)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Primary Outcome: Change From Baseline Over Time in Reported Degree of Interference With Daily Function Caused by Vomiting, as Assessed Through Use of the NCI PRO-CTCAE
Description: as for outcome 4
Time Frame: Baseline, Day 1 of each treatment cycle (1 cycle is 28 days), and at study drug discontinuation (up to 2 years)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Primary Outcome: Change From Baseline Over Time in Overall Score for Vomiting, as Assessed Through Use of the NCI PRO-CTCAE
Description: as for outcome 4
Time Frame: Baseline, Day 1 of each treatment cycle (1 cycle is 28 days), and at study drug discontinuation (up to 2 years)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Primary Outcome: Number of Participants Reporting Presence or Absence of Diarrhea Over Time, as Assessed Through Use of the NCI PRO-CTCAE Over Time
Description: as for outcome 4
Time Frame: Day 1 of each treatment cycle (1 cycle is 28 days) and at study drug discontinuation (up to 2 years)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Primary Outcome: Change From Baseline in Reported Frequency of Diarrhea Over Time, as Assessed Through Use of the NCI PRO-CTCAE
Description: as for outcome 4
Time Frame: Baseline, Day 1 of each treatment cycle (1 cycle is 28 days), and at study drug discontinuation (up to 2 years)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Primary Outcome: Change From Baseline in Reported Severity of Diarrhea Over Time, as Assessed Through Use of the NCI PRO-CTCAE
Description: as for outcome 4
Time Frame: Baseline, Day 1 of each treatment cycle (1 cycle is 28 days), and at study drug discontinuation (up to 2 years)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Primary Outcome: Change From Baseline in Reported Degree of Interference With Daily Function Caused by Diarrhea Over Time, as Assessed Through Use of the NCI PRO-CTCAE
Description: as for outcome 4
Time Frame: Baseline, Day 1 of each treatment cycle (1 cycle is 28 days), and at study drug discontinuation (up to 2 years)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

18. Primary Outcome: Change From Baseline in Overall Score for Diarrhea Over Time, as Assessed Through Use of the NCI PRO-CTCAE
Description: as for outcome 4
Time Frame: Baseline, Day 1 of each treatment cycle (1 cycle is 28 days), and at study drug discontinuation (up to 2 years)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

19. Primary Outcome: Number of Participants, Per ELN Categories, With a Complete Remission (CR) at the End of Induction Treatment, Among Those Treated at the Recommended Phase 2 Dose
Description: Sponsor's decision to prematurely terminate the study was made at the end of the Phase 1. This decision was not based on safety concerns, but rather due to the overall company strategy about the adult AML. Therefore this outcome measure was not conducted and no data available to report.
Time Frame: At the end of induction treatment (up to 2 cycles; 1 cycle is 28 days)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

20. Secondary Outcome: Dose Escalation and Expansion Phases: Percentage of Participants With a CR, Complete Remission With Incomplete Blood Count Recovery (CRi), or Complete Remission With Incomplete Platelet Count Recovery (CRp) at the End of Induction Treatment
Description: as for outcome 4
Time Frame: At the end of induction treatment (up to 2 cycles; 1 cycle is 28 days)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

21. Secondary Outcome: Dose Escalation and Expansion Phases: Percentage of Participants With a CR or Complete Remission With Partial Hematologic Recovery (CRh) at the End of Induction Treatment
Description: Sponsor's decision to prematurely terminate the study was made at the end of the Phase 1. The planned Phase 2 was not initiated. This decision was not based on safety concerns, but rather due to the overall company strategy about the adult AML. Therefore this outcome measure was not conducted and no data available to report.
Time Frame: At the end of induction treatment (up to 2 cycles; 1 cycle is 28 days)
Population: ITT Population. Analyzed population was the number of participants in Cohorts 1-3 from whom evaluable data were obtained. The Postconsidaltion cohort involved the participants in maintenance and were excluded.
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

22. Secondary Outcome: Dose-Escalation and Expansion Phases: Percentage of Participants With a Negative Minimal Residual Disease (MRD) Status at the End of Induction Treatment
Description: as for outcome 21
Time Frame: At the end of induction treatment (up to 2 cycles; 1 cycle is 28 days)
Population: as for outcome 21
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

23. Secondary Outcome: Post-Consolidation Phase: Percentage of Participants Converting From MRD-Positive to MRD-Negative Status at Any Time During Treatment
Description: as for outcome 4
Time Frame: At the end of maintenance treatment (12 cycles, 1 cycle is 28 days)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

24. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants in Event-Free Survival
Description: as for outcome 4
Time Frame: Up to 5 years
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

25. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants in Overall Survival
Description: as for outcome 4
Time Frame: Up to 5 years
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

26. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants in Relapse-Free Survival in Those Who Achieve Remission (CR, CRi, CRp, or CRh)
Description: as for outcome 4
Time Frame: Up to 5 years
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

27. Secondary Outcome: Change From Baseline Over Time in the Participant-Reported Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Questionnaire Total Score
Description: as for outcome 4
Time Frame: Baseline, Day 1 of each cycle of induction and consolidation (1 cycle is 28 days), every 3 months starting at Cycle 1 of maintenance, and at study drug discontinuation (up to 2 years)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

28. Secondary Outcome: Change From Baseline Over Time in Physical Function Scale Score of the Participant-Reported European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire, Core 30 (EORTC QLQ-C30)
Description: as for outcome 4
Time Frame: Baseline, Day 1 of first induction cycle only, Day 1 of each subsequent treatment cycle (1 cycle is 28 days), and at study drug discontinuation (up to 2 years)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

29. Secondary Outcome: Change From Baseline Over Time in Role Function Scale Score of the Participant-Reported EORTC QLQ-C30
Description: as for outcome 4
Time Frame: as for outcome 28
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

30. Secondary Outcome: Change From Baseline Over Time in Global Health Status/Quality of Life Scale Score of the Participant-Reported EORTC QLQ-C30
Description: as for outcome 4
Time Frame: as for outcome 28
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

31. Secondary Outcome: Change From Baseline Over Time in Headache Symptom Score of the Participant-Reported European Organisation for Research and Treatment of Cancer (EORTC) Item Library Questionnaire
Description: as for outcome 4
Time Frame: as for outcome 27
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

32. Secondary Outcome: Change From Baseline Over Time in Dizziness Symptom Score of the Participant-Reported EORTC Item Library Questionnaire
Description: The Sponsor decided not to continue the study based on the overall Company strategy in AML. Due to the limited The sponsor decided not to continue the study based on the overall Company strategy in AML. Although data were collected, the small sample size and insufficient follow up rendered any analysis scientifically meaningless. As a consequence, no data were analyzed and this outcome measure was not conducted
Time Frame: as for outcome 27
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

33. Secondary Outcome: Change From Baseline Over Time in Bruising Symptom Score of the Participant-Reported EORTC Item Library Questionnaire
Description: as for outcome 4
Time Frame: as for outcome 27
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

34. Secondary Outcome: Change From Baseline Over Time in the European Quality of Life 5-Dimension, 5-Level Questionnaire (EQ-5D-5L) Index Utility Score
Description: as for outcome 4
Time Frame: Baseline, Day 1 of first induction cycle only, Day 1 of all cycles of consolidation (1 cycle is 28 days), every 3 months starting at Cycle 1 of maintenance, and at study drug discontinuation (up to 2 years)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

35. Secondary Outcome: Change From Baseline Over Time in the EQ-5D-5L Visual Analogue Scale (VAS) Score
Description: as for outcome 4
Time Frame: as for outcome 34
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

36. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) of Idasanutlin
Description: as for outcome 4
Time Frame: Pre-dose and at predefined intervals post-dose on Days 1, 3, and 5 of induction Cycle 1; Days 1 and 5 of consolidation Cycle 1; and Days 1 and 5 of maintenance Cycle 1 (1 cycle is 28 days)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

37. Secondary Outcome: AUC of Cytarabine
Description: as for outcome 4
Time Frame: Pre-dose and at predefined intervals post-dose on Days 1, 3, and 5 of induction Cycle 1; and Days 1 and 5 of consolidation Cycle 1 (1 cycle is 28 days)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

38. Secondary Outcome: AUC of Daunorubicin
Description: as for outcome 4
Time Frame: Pre-dose and at predefined intervals post-dose on Days 1, 3, and 5 of induction Cycle 1 (1 cycle is 28 days)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

39. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Idasanutlin
Description: as for outcome 4
Time Frame: as for outcome 36
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

40. Secondary Outcome: Cmax of Cytarabine
Description: as for outcome 4
Time Frame: as for outcome 37
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

41. Secondary Outcome: Cmax of Daunorubicin
Description: as for outcome 4
Time Frame: Pre-dose and at predefined intervals post-dose on Days 1, 3, and 5 of induction Cycle 1 (1 cycle is 28 days)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

42. Secondary Outcome: Total Clearance (CL) of Idasanutlin
Description: as for outcome 4
Time Frame: as for outcome 36
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

43. Secondary Outcome: CL of Cytarabine
Description: as for outcome 4
Time Frame: as for outcome 37
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

44. Secondary Outcome: CL of Daunorubicin
Description: as for outcome 4
Time Frame: Pre-dose and at predefined intervals post-dose on Days 1, 3, and 5 of induction Cycle 1 (1 cycle is 28 days)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

45. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Idasanutlin
Description: as for outcome 4
Time Frame: as for outcome 36
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

46. Secondary Outcome: Vss of Cytarabine
Description: as for outcome 4
Time Frame: as for outcome 37
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

47. Secondary Outcome: Vss of Daunorubicin
Description: as for outcome 4
Time Frame: Pre-dose and at predefined intervals post-dose on Days 1, 3, and 5 of induction Cycle 1 (1 cycle is 28 days)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

48. Secondary Outcome: Terminal Half-Life (t1/2) of Idasanutlin
Description: as for outcome 4
Time Frame: as for outcome 36
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

49. Secondary Outcome: t1/2 of Cytarabine
Description: as for outcome 4
Time Frame: as for outcome 37
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

50. Secondary Outcome: t1/2 of Daunorubicin
Description: as for outcome 4
Time Frame: Pre-dose and at predefined intervals post-dose on Days 1, 3, and 5 of induction Cycle 1 (1 cycle is 28 days)
Population: as for outcome 4
Arm/Group | Dose-Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | Post Consolidation Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline up to 28 days after the last study treatment depending on the stage of the study. The study was prematurely terminated. The last participant's last treatment was at Induction Cycle 1 Day 7.
Description: Treatment and SFU
Groups:
- DOSE ESCALATION COHORT 1: For induction, participants will be treated with idasanutlin plus cytarabine and daunorubicin. At the investigator's discretion for consolidation, either participants will be treated with idasanutlin and cytarabine or they will undergo Allo-HSCT. For maintenance, participants will be treated with single-agent idasanutlin of 200 mg
- POST CONSOLIDATION PHASE COHORT: Participants who are idasanutlin treatment-naive, had received induction and chemotherapy consolidation for AML outside of the study, and were in minimal residual disease (MRD)-positive remission after induction will be enrolled in this cohort to receive maintenance treatment with single-agent idasanutlin of 150 mg
Arm/Group | DOSE ESCALATION COHORT 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3 | POST CONSOLIDATION PHASE COHORT
All-Cause Mortality (participants affected / at risk) | 2/4 | 1/9 | 0/6 | 1/4
Serious Adverse Events (participants affected / at risk) | 3/4 | 4/9 | 2/6 | 1/4
Other Adverse Events (participants affected / at risk) | 4/4 | 9/9 | 6/6 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOSE ESCALATION COHORT 1 (N=4) | Dose Escalation Cohort 2 (N=9) | Dose Escalation Cohort 3 (N=6) | POST CONSOLIDATION PHASE COHORT (N=4)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3) | 2 (5) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOSE ESCALATION COHORT 1 (N=4) | Dose Escalation Cohort 2 (N=9) | Dose Escalation Cohort 3 (N=6) | POST CONSOLIDATION PHASE COHORT (N=4)
Anaemia (Blood and lymphatic system disorders) | 2 (5) | 4 (5) | 2 (4) | 1 (10)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4) | 8 (11) | 4 (4) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (7) | 0 (0) | 0 (0) | 3 (14)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (17)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (8) | 4 (5) | 3 (3) | 4 (9)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (4) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ear swelling (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Papilloedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 9 (14) | 5 (9) | 3 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 8 (11) | 4 (5) | 4 (6)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (5) | 2 (3) | 3 (3) | 0 (0)
Tongue discolouration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 4 (5) | 3 (4) | 2 (3)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (5)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Face oedema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 3 (3) | 3 (4) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Mucosal inflammation (General disorders) | 1 (1) | 6 (6) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 3 (3) | 5 (7) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 1 (3) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Physical deconditioning (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacillus bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Bacteroides bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Scrotal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 4 (9) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Blood count abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactic acid increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 2 (8) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 2 (4) | 1 (3)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 2 (5) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (4)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (15) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (7) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (8) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 4 (11) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (6) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 3 (5) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (4) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 3 (4) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukoplakia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Onychalgia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (5) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 4 (5) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 4 (4) | 1 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxic erythema of chemotherapy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 3 (5) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/35/NCT03850535/Prot_SAP_000.pdf